CLINICAL TRIAL: NCT02471014
Title: The Effect of Obesity on Immune Responses to Pneumococcal Polysaccharide Vaccine, ROVE Study
Brief Title: Effect of Obesity on Immune Response to Pneumovax 23
Acronym: ROVE
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201401069
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Obesity
Keywords: Pneumovax23; Obesity
MeSH Terms: conditions — Obesity | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Pneumococcal Vaccines; Hematologic Tests; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese Individuals: Participants in this group will receive one 0.5mL Pneumovax23 intramuscular vaccine at baseline, four questionnaires administered at baseline, and one 50mL blood draw at baseline and one 50mL blood draw up to 6 weeks later.
  Interventions: Drug: Pneumovax 23; Other: Blood tests; Other: Questionnaires
- Normal Individuals: Participants in this group will receive one 0.5mL Pneumovax23 intramuscular vaccine at baseline, four questionnaires administered at baseline, and one 50mL blood draw at baseline and one 50mL blood draw up to 6 weeks later.
  Interventions: Drug: Pneumovax 23; Other: Blood tests; Other: Questionnaires

INTERVENTIONS:
Drug: Pneumovax 23 — All participants will receive a single 0.5 mL Pneumovax 23 intramuscular vaccine at baseline.
  Other Names: pneumococcal polysaccharide vaccine
Other: Blood tests — All participants will have two 50 milliliter blood draws: at baseline and up to 6 weeks later.
Other: Questionnaires — All participants will answer the following questionnaires:
  UCLA Loneliness Scale Questionnaire will be used to measure a difference between the groups.
  Perceived Stress Scale-10 Questionnaire will be used to measure a difference between the groups.
  Interpersonal Support Evaluation List-12 will be used to measure a difference between the groups Life Orientation Test-Revised will be used to measure a difference between the groups.

SUMMARY:
Pneumococcal infections are a leading cause of adult and childhood hospitalization and death. It has been shown that obese individuals are at higher risk for this bacterial infection. As a result, investigators will vaccinate obese individuals to see if they are offered the same level of protection from the vaccine as normal-weight individuals. The vaccine used for this particular bacterial infection is called Pneumovax 23.

The purpose of this study is to compare how body mass index affects protection that the vaccine provides against these bacteria.

Primary Hypothesis: Levels of protection from the vaccine are no different in pre- and post- vaccination in healthy BMI individuals and obese individuals.

DETAILED DESCRIPTION:
Study Participants: For this study, the investigators will recruit 56 participants separated into two groups. Group 1 will enroll 23 individuals with a BMI between 22 and 25. Group 2 will enroll 23 obese individuals. Study participants will be between the ages of 18-35 and in good health.

Pre-Screening: Basic eligibility will first be determined by phone or through a questionnaire. The investigators will acquire weight and height information to calculate BMI, as well as ask about any chronic health problems. At the end of the pre-screening, an email address will be requested in order to email a copy of the consent form for the participant to review before the first visit, during which the consent form will be reviewed with the participant and any questions addressed. A cell phone number will also be requested to text participant reminders the night before their appointments (visit 1 and visit 2). If the participant declines a reminder text, a reminder phone call will be set-up.

Screening: During the in-person screening, the investigators will ask several questions. Participants with chronic health problems (significant vascular disease, hepatitis, renal disease, diabetes, immunodeficiency) will be excluded. Individuals already immunized with Pneumovax23 or Prevnar (another vaccine that protects against pneumococcal infection) will also be excluded. A pregnancy test will be given to females to exclude pregnant individuals. An HbA1C (finger prick to get a drop of blood) will also be performed to exclude participants with high blood sugar levels. Physical exams will be performed and vitals will be taken on participants who pass the initial screening to help assess health.

Questionnaires will also be given at the first visit to assess stress, which has been shown to affect the ability to protect against infection.

Study Visits: All participants will receive a Pneumovax 23 vaccine, questionnaires, physical exams, and undergo 2 blood draws.

Part of the blood will be sent to a research laboratory for gene analysis. This will help us determine if certain genetic markers explain individual differences in Pneumovax 23 efficacy.

ELIGIBILITY:
Inclusion Criteria:

Control group

* aged 18-35
* BMIs between 22-25kg/m2, Obese group
* Aged 18 - 35
* BMIs greater than 30kg/m2, and
* waist to hip ratio of at least 0.9 in males and at least 0.85 in females

Exclusion Criteria:

* Pregnancy: Pregnant, Planning to become pregnant, or Breastfeeding
* Diabetes mellitus (A1C> 6.5%): Diagnosed with diabetes
* Abnormal CMP and CBC values as determined by the Principal Investigator.
* Inability to fast for 8 hours prior to the initial blood draw
* Immunization: Immunized with Pneumovax 23, or Immunized with Prevnar
* Medications:Currently taking any of the following medications or within the 4 weeks of study:

  i. Immunosuppressive drugs or chemotherapeutic agents such as azathioprine, mycophenolate mofetil, TNF inhibitors, cyclosporine, methotrexate, leflunomide, cyclophosphamide, sulfasalazine, antimalarial drugs, chlorambucil, nitrogen mustard

ii. Steroids such as prednisone, cortisone, hydrocortisone

iii. Antidiabetic drugs such as metformin, insulin, glipizide, meglitinide, sulfonylurea, glimepiride, repaglinide, nateglinide

* History of clinical illness (exclusion during clinic)

  1. Pneumonia or Previously had Pneumonia
  2. Low blood pressure or Experienced dizzy spells
  3. Significant cardiovascular disease:Recently hospitalizations deemed significant at the discretion of the Principal Investigator, or History of heart attack, or History of stroke
  4. Spleen, Splenectomy, or Damage to spleen
  5. Lung Disease or History of lung disease
  6. Kidney disease, Blood in urine, or Protein in urine
  7. Liver disease, Previous or current liver diseases such as hepatitis A, B, or C, liver cirrhosis, or autoimmune hepatitis, or Elevated AST/ALT lab test
  8. Leukopenias
  9. Hemoglobinopathies, History of sickle cell disease, or thalassemia
  10. HIV/AIDS, or a history of HIV infection
  11. Recreational IV drug use, or Intravenous drug injection predisposes users to infections, such as human immunodeficiency virus, that may alter the immune system and therefore affect the immunoglobulin response to Pneumovax23.
  12. History of IV-drug use, or IV drug use is a risk factor for HIV infection, which may change the immune response to Pneumovax 23.
  13. History of idiopathic thrombocytopenic purpura
  14. History of chronic inflammatory diseases such as rheumatoid arthritis or chronic granulomatous disease
  15. Autoimmune disease
  16. Immunodeficiencies: neutropenia, common variable immune deficiency, Bruton's X-linked agammaglobulinemia; SCID; Selective IgA deficiency; Wiskott-Aldrich Syndrome; Ataxia Telangiectasia; DiGeorge Syndrome; Chronic Granulomatous Disease; Hyper IgE Syndrome; Complement deficiencies
* Weight

  1. Planning on losing weight within the time frame of the study
  2. Have experienced excessive weight loss or gain within two months prior to the study
  3. Planning to undergo liposuction, gastric bypass, stomach stapling, whipple procedure, or reconstructive surgery involving transplantation of adipose tissue within the study period
  4. Bodybuilder or someone who takes part in excessive weight training
* Allergy

  1. Any severe side effects from vaccines
  2. Allergic reaction to phenol
* Medications/Supplementations

  1. Taking any antioxidant supplements (EmergenC)
  2. Unable to refrain from antioxidant supplements throughout the duration of the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Area County Adults residents with a diagnosis of Obesity who are otherwise healthy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Brantly, MD, Principal Investigator — Professor of Medicine & Chief, Division of Pulmonary, Critical Care & Sleep Medicine
Locations (1):
- Uf Ctsi Crc, Gainesville, Florida, United States

REFERENCES:
- [Result] Sebastian M, Hsiao CJ, Futch HS, Eisinger RS, Dumeny L, Patel S, Gobena M, Katikaneni DS, Cohen J, Carpenter AM, Spiryda L, Heldermon CD, Jin L, Brantly ML. Obesity and STING1 genotype associate with 23-valent pneumococcal vaccination efficacy. JCI Insight. 2020 May 7;5(9):e136141. doi: 10.1172/jci.insight.136141. PMID 32376795

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 56 consented. 6 participants failed secondary screening during the first visit.
Groups:
- Obese Individuals; Normal Individuals: Participants in this group will receive one 0.5mL Pneumovax23 intramuscular vaccine at baseline, four questionnaires administered at baseline, and one 50mL blood draw at baseline and one 50mL blood draw up to 6 weeks later.
  Pneumovax 23: All participants will receive a single 0.5 mL Pneumovax 23 intramuscular vaccine at baseline.
  Blood tests: All participants will have two 50 milliliter blood draws: at baseline and up to 6 weeks later.
  Questionnaires: All participants will answer the following questionnaires:
  UCLA Loneliness Scale Questionnaire will be used to measure a difference between the groups.
  Perceived Stress Scale-10 Questionnaire will be used to measure a difference between the groups.
  Interpersonal Support Evaluation List-12 will be used to measure a difference between the groups Life Orientation Test-Revised will be used to measure a difference between the groups.
Period: Overall Study
Arm/Group | Obese Individuals | Normal Individuals
Started | 25 | 25
Completed | 23 | 23
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: The baseline population is the same.
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese Individuals | Normal Individuals | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (5.32) | 23.0 (3.08) | 26.0 (5.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 0 | 5
  White | 12 | 17 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Anti-pneumococcal Antibodies Between the Groups
Description: IgG antibody titers specific for each serotype in Pneumovax 23 (i.e. 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19F, 19A, 20, 22F, 23F, and 33F) will be analyzed.
Time Frame: Changes in baseline and up to 6 weeks
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Obese Individuals | Normal Individuals
Number analyzed (Participants) | 23 | 23
titer | 34.1 (3.51) | 19.8 (1.52)

2. Secondary Outcome: UCLA Loneliness Scale Questionnaire Will be Used to Measure a Difference Between the Groups.
Description: The UCLA loneliness scale is a 20-item questionnaire, on a scale of 0-3 for each question. This questionnaire measures subjective feelings of loneliness and social isolation. Final score of 0 reflects no loneliness and 60 reflects the maximum amount of loneliness.
Time Frame: Baseline
Reporting Status: Not Posted

3. Secondary Outcome: Perceived Stress Scale-10 Questionnaire Will be Used to Measure a Difference Between the Groups.
Description: The Perceived Stress Scale-10 is a 10-item questionnaire assessing how stressful participants perceive their lives to be. Each question is assessed on a scale of 0 to 4. Final score of 0 reflects no stress and 40 indicates maximum amount of stress.
Time Frame: Baseline
Reporting Status: Not Posted

4. Secondary Outcome: Interpersonal Support Evaluation List-12 Will be Used to Measure a Difference Between the Groups
Description: The Interpersonal Support Evaluation List-12, a 12-item questionnaire that measures perceived social support along 3 dimensions: appraisal support (availability of someone to talk to), belonging support (availability of people to do things with), and tangible support (e.g. material aid). This is measured on a scale of 0 to 36. The greater the number the greater perceived support.
Time Frame: Baseline
Reporting Status: Not Posted

5. Secondary Outcome: Life Orientation Test-Revised Will be Used to Measure a Difference Between the Groups.
Description: The Life Orientation Test-Revised, a 10-item scale measuring optimism versus pessimism along a continuous scale; a higher score indicates more optimism. The lowest score is 0 and the highest is 24.
Time Frame: Baseline
Reporting Status: Not Posted

6. Secondary Outcome: Genetic Analysis
Description: A small amount of blood will be sent to a research laboratory for an analysis of genetic markers Specifically, we will be analyzing the the stimulator of interferon genes (STING). This will help us determine if this gene, which has been previously thought to contribute to Pneumovax efficacy, helps explain individual differences in immune response.
Time Frame: Test to be performed in a research laboratory after Visits are completed
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4-6 weeks
Description: No subjects experienced serious adverse events.
Arm/Group | Obese Individuals | Normal Individuals
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT02471014/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT02471014/SAP_001.pdf